CLINICAL TRIAL: NCT00281216
Title: Innate and Adaptive Immunity in COPD Exacerbations: Prospective Cohort Study
Brief Title: Innate and Adaptive Immunity in Individuals Experiencing Chronic Obstructive Pulmonary Disease Exacerbations
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey L. Curtis, Professor of Internal Medicine (Pulmonary & Critical Care Medicine Division), University of Michigan
Other Study IDs: 1324; R01HL082480 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, sputum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether there is a statistical association between the changes from baseline in the levels of two cytokines interleukin (IL)-17A and IL-6 in the sputum of patients with chronic obstructive pulmonary disease (COPD) and the severity of acute exacerbations of COPD (AE-COPD). These sputum cytokine levels are taken as measures of the adaptive immune response (IL-17A) and the innate immune response (IL-6), respectively. Sputum will be collected either spontaneously or will be obtained by induction; cytokine levels will be measured by ELISA. The primary analysis, comparisons of sputum cytokine levels between clinical states, will be done using random effects modeling.

DETAILED DESCRIPTION:
BACKGROUND:

COPD is one of the most pressing healthcare problems facing our nation. AE-COPD is responsible for the bulk of healthcare costs and much of the morbidity and decline in health status among individuals with this common disease. The lack of accepted animal models of AE-COPD necessitates novel approaches using human samples. Advances in the understanding of the pathogenesis have been slowed, in part, due to controversy as to how exacerbations should be defined. The prevailing paradigm has defined AE-COPD as event-based. Such definitions clearly identify groups of patients with accelerated loss of pulmonary function and increased mortality. However, limited data show that symptom-based definitions of AE-COPD also capture episodes inducing significant morbidity and functional decline, and hence of concern to patients. Fundamental mechanisms are lacking to explain AE-COPD defined by either means.

Controversy also surrounds triggers of AE-COPD. Bacteria and viruses are involved in some episodes, but the relative importance of each is intertwined with disputes over the definition of AE-COPD. Progress at linking specific pathogens to molecular pathogenesis has been slow, both due to their diversity, and to the high rates of bacterial colonization of patients with COPD, even in the stable state. Moreover, in many AE-COPD cases, no pathogen can be identified. Without negating the value of analyzing infections with specific species of pathogens, it appears that progress in molecular pathogenesis could be accelerated by focusing on unifying features of the pulmonary immune response during AE-COPD.

DESIGN NARRATIVE:

A prospective patient cohort will be studied extensively physiologically, functionally, and immunologically upon enrollment while in the stable state. As part of the study, participants will be trained in the use of peak flow meters, so that they can record daily first morning peak expiratory flow rates (PEFR). To confirm the range of fluctuations in their basal state, participants will be then be followed at three-month intervals for face-to-face interviews and more limited physiological and functional testing described below. Participants will also be reminded at each scheduled visit to contact the study coordinator when they feel that an AE-COPD may be present. If they do contact the study coordinator, they will be evaluated at one of the study sites within 48 hours.

A diagnosis of AE-COPD will incorporate a modification of the definition used by the COPD Clinical Research Network (CCRN). The diagnosis will be made in one of two ways: severe AE-COPD will be defined as a change in respiratory symptoms above the participant's baseline measurements plus evaluation in the emergency room (ER) or requiring hospitalization; or mild-to-moderate AE-COPD will be defined as a change in respiratory symptoms above the participant's baseline measurements and requiring a change in therapy (addition of either antibiotics, oral steroids, or both), but without evaluation in the ER or hospitalization. In the latter case, therapy could be changed either at the advice of the patient's own caregivers or a study physician based on clinical judgment, or could be self-initiated in the case of participants authorized to do so by their caregiver. A concerted effort will be made to capture these milder AE-COPD during both winter and non-winter seasons.

Upon enrolling participants, the following will be performed: review of medical history; review of demographic and smoking history; physical examination, blood and sputum collection; six-minute walk test; and questionnaires to assess shortness of breath (MMRC and University of California San Diego SOBQ), sputum production (modified Chronic Bronchitis Symptom Questionnaire), health status (SF-36 and St. George's Respiratory Questionnaire), and psychological traits (Hospital Anxiety/Depression Score, Illness Perception Questionnaire, Coping Index, and an individualized 30-minute clinical interview via telephone).

Participants will attend study visits every 3 months to review symptoms. During an AE-COPD (episode of acute bronchitis), sputum and blood will be collected, and a five-symptom questionnaire will be filled out.

Subjects are reimbursed $25 per scheduled visit and $50 per unscheduled visit (at the time of perceived exacerbation) to help defray travel expenses.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD (following American Thoracic Society guidelines) and/or chronic bronchitis
* Forced Expiratory Volume in 1 second of less than 70% predicted value after bronchodilator
* Current or former smokers with more than 20 pack-years
* Daily productive cough for 3 months of the year for 2 consecutive years
* At least one AE-COPD requiring medical attention in each year for the previous 3 years
* Willingness to participate in follow-up studies defined in the protocol

Exclusion criteria:

* Unstable cardiovascular disease
* Other systemic disease in which survival of more than 2 years is unlikely
* Mental incompetence or active psychiatric illness
* Currently taking more than 20 mg/day of Prednisone
* Participation in another experimental protocol within 6 weeks of study entry
* Asthma
* Cystic fibrosis
* Clinically significant bronchiectasis
* Lung cancer
* Other inflammatory or fibrotic lung disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruited from pulmonary and general medicine clinics
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Curtis, Study Chair — University of Michigan at Ann Arbor
Locations (1):
- University of Michigan at Ann Arbor, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Freeman CM, Curtis JL, Chensue SW. CC chemokine receptor 5 and CXC chemokine receptor 6 expression by lung CD8+ cells correlates with chronic obstructive pulmonary disease severity. Am J Pathol. 2007 Sep;171(3):767-76. doi: 10.2353/ajpath.2007.061177. Epub 2007 Jul 19. PMID 17640964
- [Background] Curtis JL, Freeman CM, Hogg JC. The immunopathogenesis of chronic obstructive pulmonary disease: insights from recent research. Proc Am Thorac Soc. 2007 Oct 1;4(7):512-21. doi: 10.1513/pats.200701-002FM. PMID 17878463
- [Result] Freeman CM, Martinez FJ, Han MK, Washko GR Jr, McCubbrey AL, Chensue SW, Arenberg DA, Meldrum CA, McCloskey L, Curtis JL. Lung CD8+ T cells in COPD have increased expression of bacterial TLRs. Respir Res. 2013 Feb 1;14(1):13. doi: 10.1186/1465-9921-14-13. PMID 23374856
- [Result] Freeman CM, Han MK, Martinez FJ, Murray S, Liu LX, Chensue SW, Polak TJ, Sonstein J, Todt JC, Ames TM, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Cytotoxic potential of lung CD8(+) T cells increases with chronic obstructive pulmonary disease severity and with in vitro stimulation by IL-18 or IL-15. J Immunol. 2010 Jun 1;184(11):6504-13. doi: 10.4049/jimmunol.1000006. Epub 2010 Apr 28. PMID 20427767
- [Result] Freeman CM, Martinez FJ, Han MK, Ames TM, Chensue SW, Todt JC, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Lung dendritic cell expression of maturation molecules increases with worsening chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Dec 15;180(12):1179-88. doi: 10.1164/rccm.200904-0552OC. Epub 2009 Sep 3. PMID 19729666
- [Result] Freeman CM, Martinez CH, Todt JC, Martinez FJ, Han MK, Thompson DL, McCloskey L, Curtis JL. Acute exacerbations of chronic obstructive pulmonary disease are associated with decreased CD4+ & CD8+ T cells and increased growth & differentiation factor-15 (GDF-15) in peripheral blood. Respir Res. 2015 Aug 5;16(1):94. doi: 10.1186/s12931-015-0251-1. PMID 26243260
- See also: Curtis Laboratory — http://www.copdfoundation.org/
- See also: COPD Foundation — http://www.copdfoundation.org/